CLINICAL TRIAL: NCT00008294
Title: A Phase I Study Of Hepatic Arterial Infusion With Floxuridine And Dexamethasone In Combination With Intravenous Oxaliplatin Plus 5-Fluorouracil And Leucovorin In Patients With Unresectable Hepatic Metastases From Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Unresectable Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-009; P30CA008748 (NIH); MSKCC-00009; NCI-G00-1896
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Dexamethasone; Floxuridine; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: dexamethasone
Drug: floxuridine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Cryosurgery kills cancer cells by freezing them. Combining more than one chemotherapy drug with cryosurgery and giving drugs in different ways may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of intrahepatic and intravenous combination chemotherapy with or without cryosurgery in treating unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oxaliplatin and fluorouracil when given with leucovorin calcium and hepatic intra-arterial floxuridine and dexamethasone with or without cryosurgery (group I cryosurgery closed to accrual as of 10/13/03) in patients with unresectable liver metastases from colorectal cancer.
* Determine, preliminarily, the anti-tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of oxaliplatin and fluorouracil. Patients are assigned to one of two treatment groups. (Group I closed to accrual as of 10/13/03.)

* Group I (closed to accrual as of 10/13/03): Patients with no more than 8 hepatic metastases and no metastases greater than 5 cm in diameter undergo cryosurgery prior to chemotherapy. Chemotherapy is delayed for at least 4 weeks after cryosurgery.
* Group II: Patients with more than 8 hepatic metastases or at least one metastases greater than 5 cm in diameter do not undergo cryosurgery prior to chemotherapy.

Beginning 2 weeks after pump placement surgery, all patients receive floxuridine and dexamethasone by hepatic intra-arterial infusion continuously on days 1-14; oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on days 15 and 29; and fluorouracil IV continuously over 48 hours on days 15-16 and 29-30. Courses repeat every 36 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and fluorouracil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 4-72 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum with unresectable liver metastases that comprise less than 70% of liver parenchyma

  * No extrahepatic disease
* No ascites

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* No hepatic encephalopathy

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No obstruction of gastrointestinal tract or genitourinary tract
* No symptomatic peripheral sensory neuropathy
* No active infection
* No other malignancy except resectable primary colorectal carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior floxuridine
* If undergoing cryosurgery (group I cryosurgery closed to accrual as of 10/13/03), must have received one of the following:

  * Systemic chemotherapy for metastatic disease
  * Adjuvant therapy within the past 6 months comprising fluorouracil with or without levamisole for resected primary colorectal carcinoma
  * Adjuvant therapy within the past 12 months comprising fluorouracil and leucovorin calcium with or without levamisole for resected primary colorectal carcinoma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to liver

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Kemeny, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kemeny N, Capanu M, D'Angelica M, Jarnagin W, Haviland D, Dematteo R, Fong Y. Phase I trial of adjuvant hepatic arterial infusion (HAI) with floxuridine (FUDR) and dexamethasone plus systemic oxaliplatin, 5-fluorouracil and leucovorin in patients with resected liver metastases from colorectal cancer. Ann Oncol. 2009 Jul;20(7):1236-41. doi: 10.1093/annonc/mdn769. Epub 2009 Feb 20. PMID 19233901
- [Result] Kemeny N, Jarnagin W, Paty P, Gonen M, Schwartz L, Morse M, Leonard G, D'Angelica M, DeMatteo R, Blumgart L, Fong Y. Phase I trial of systemic oxaliplatin combination chemotherapy with hepatic arterial infusion in patients with unresectable liver metastases from colorectal cancer. J Clin Oncol. 2005 Aug 1;23(22):4888-96. doi: 10.1200/JCO.2005.07.100. Epub 2005 Jul 11. PMID 16009951